CLINICAL TRIAL: NCT04067362
Title: The Effects of 2 Inulin Sources on Satiety and Gastrointestinal Tolerance
Brief Title: Chicory Fiber Effect on Satiety and GI Tolerance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY000179126
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no fiber (Placebo Comparator): Breakfast with hot chocolate with no fiber
  Interventions: Other: food containing dietary fiber
- chicory root flour (Experimental): Breakfast with hot chocolate with chicory root flour
  Interventions: Other: food containing dietary fiber
- chicory root fiber supplement (Experimental): Breakfast with hot chocolate with chicory root fiber supplement
  Interventions: Other: food containing dietary fiber

INTERVENTIONS:
Other: food containing dietary fiber — commercially available chicory root flour and chicory root fiber

SUMMARY:
The investigators are comparing 2 fiber treatments to a fiber free treatment for acute satiety and GI response.

DETAILED DESCRIPTION:
The investigators are measuring satiety and GI response after subjects consume 3 acute breakfast meals: 1. fiber-free control; 2. chicory root flour containing inulin; 3. inulin fiber supplement. After breakfast, subjects will complete subjective satiety instruments and describe any GI symptoms.

ELIGIBILITY:
Inclusion Criteria:

no food allergies; healthy; willing to consume breakfast in laboratory setting; usual low fiber diet;

Exclusion Criteria:

smokers, taking dietary supplements containing fiber

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
satiety | 2 hours
  subjective instrument to assess how full you feel

SECONDARY OUTCOMES:
Gastrointestinal response | 24 hours
  subjective description of any GI symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No